CLINICAL TRIAL: NCT00304837
Title: VEGF Gene Transfer for Critical Limb Ischemia
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Losordo, Douglas, M.D. (Individual)
Allocation: Randomized | Model: Crossover | Masking: Double
Other Study IDs: BB-IND 11948
Record Dates: First submitted 2006-03-16; First posted 2006-03-20 (Estimated); Last update posted 2010-10-19 (Estimated); Status verified 2008-04

CONDITIONS: Critical Limb Ischemia; Ischemia; Leg Ulcer
Keywords: Nonhealing leg ulcers; Ischemic rest pain
MeSH Terms: conditions — Chronic Limb-Threatening Ischemia; Ischemia; Leg Ulcer

INTERVENTIONS:
Genetic: pVGI.1 (VEGF-2)

SUMMARY:
The purpose of this gene therapy study is to evaluate the safety and efficacy of intramuscular gene transfer using Vascular Endothelial Growth Factor (VEGF) or placebo in patients with moderate to high-risk Critical Limb Ischemia (a condition in which there is poor blood circulation in the leg). This trial will assess whether VEGF improves rest pain and/or heals ulcers in the legs of patients with peripheral artery disease (blockages in leg arteries.)

VEGF is DNA, or genetic material that will be injected into the leg muscles on three separate occasions, each 2 weeks apart. Once the DNA is in the leg, it directs the cells of the artery wall to increase its production of VEGF, which has been shown to cause new blood vessels to grow. This experimental therapy is designed to grow new blood vessels around blockages in the leg arteries.

The total length of participation in this study is approximately 1 year and will require approximately 8 clinic visits within that year. Following enrollment in the study, testing may be done for cancer screening, blood work, physical exams, vascular testing and eye exams. There is no charge for any testing or office visits required by the study.

This study has been approved by the Food and Drug Administration (FDA).

ELIGIBILITY:
Inclusion Criteria:

* Be at least 21 years old
* Have critical limb ischemia
* Have severe blockages in at least one artery in the affected leg as demonstrated by an angiogram
* Have nonhealing leg ulcers and/ or have severe rest pain secondary to a severely decreased blood flow
* Agree to participate in follow-up.

Exclusion Criteria:

* Have any evidence of malignant neoplasms (other than non-melanoma skin cancer or in situ carcinoma) within the last 5 years
* Be pregnant or lactating
* Have a history of alcohol or drug abuse within 3 months of screening
* Have advanced (Rutherford Category 6) critical limb ischemia, characterized by extensive tissue loss or gangrene
* Have osteomyelitis
* Have undergone successful aortic or lower extremity surgery, angioplasty, or lumbar sympathectomy within the 2 months preceding screening
* Be a suitable candidate for surgical or endovascular revascularization in the limb in which treatment is proposed
* Subjects in whom arterial insufficiency in the lower extremity is the result of a non-atherosclerotic disorder

Min Age: 21 Years | Sex: All
Age Groups: Adult, Older Adult
Dates: Study Completion 2008-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Douglas W. Losordo, MD, Study Director — Northwestern University
Locations (3):
- United States (3):
  - Cardiology PC, Birmingham, Alabama
  - Caritas St. Elizabeth's Medical Center, Boston, Massachusetts
  - The Minneapolis Heart Institute at Abbott Northwestern Hospital, Minneapolis, Minnesota